CLINICAL TRIAL: NCT01715714
Title: Statin Recapture Therapy Before Coronary Artery Bypass Grafting
Acronym: StaRT-CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, PD Dr. Oliver J. Liakopoulos, Principal Investigator, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-1341; 2011-001795-19 (EudraCT Number); DRKS00000753 (Registry Identifier: German Clinical Trials Register (DRKS))
Record Dates: First submitted 2012-10-18; First posted 2012-10-29 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Statins; Coronary Artery Bypass Grafting; Cardiac Surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Simvastatin; Atorvastatin; Pravastatin; Fluvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin Recapture Therapy (Active Comparator): Oral statin reload of patients at 12 and 2 hours before CABG using the maximal dose of the chronically prescribed statin* on admission. (*simvastatin 80 mg, atorvastatin 80 mg, fluvastatin 80 mg or pravastatin 40 mg)
  Interventions: Drug: Statin Recapture Therapy
- Placebo (Placebo Comparator): Placebo given orally 12 hrs and 2 hrs before CABG
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Statin Recapture Therapy — Given 12h and 2h before CABG
  Other Names: Simvastatin 80 mg; Atorvastatin 80 mg; Pravastatin 40 mg; Fluvastatin 80 mg
  Arms: Statin Recapture Therapy
Drug: Placebo — Given 12h and 2h before CABG.
  Arms: Placebo

SUMMARY:
Patients with coronary artery disease requiring coronary artery bypass grafting (CABG) are at risk for postoperative complications after surgery. The StaRT-CABG trial is the first large-scale (2,630 patients) that will investigate whether an additional treatment with statins (lipid-lowering medication) in high doses before CABG surgery can reduce the incidence of major post-surgery complications including death, myocardial infarction and stroke. The StaRT-CABG trial will be recruiting patients from 8 cardiac surgery centres in Germany and is expected to provide relevant clinical data on the efficacy of this novel treatment in order to optimize the care for all patients undergoing CABG.

DETAILED DESCRIPTION:
Patients with coronary artery disease (CAD) requiring coronary artery bypass grafting (CABG) are still at significant risk for postoperative major adverse cardiocerebral events (≈15% MACCE rate), with ≈3% of patients dying within 30 days of surgery. Recent clinical evidence shows that cardioprotection in patients receiving chronic statin treatment can be further improved by a high-dose statin 'recapture' therapy given shortly before an ischemia-reperfusion sequence, resulting in a 61% risk reduction for MACE at 30 days in patients undergoing PCI. Evaluation of this novel approach in the setting of CABG seems particularly promising, as myocardial injury, surgery-related inflammation and pre-existing patients' comorbidities play a pivotal role for poor clinical outcomes after CABG that may be improved by an acute statin recapture therapy. The StaRT-CABG trial is the first large-scale (n=2,630 CABG patients), multicentre (8 cardiac surgery centres), randomised, double-blind and placebo-controlled trial that aims to test whether an acute high-dose statin recapture therapy given shortly before CABG reduces the incidence of MACCE at 30 days after surgery (composite primary outcome: all-cause mortality; non-fatal myocardial infarction and cerebrovascular events). The StaRT-CABG trial is expected to provide highly relevant clinical data on the efficacy of this novel therapeutic approach in order to optimize the care for all CAD patients undergoing CABG with broad clinical implications on current clinical practice and existing guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on chronic statin treatment (>30 days) scheduled for isolated CABG, including on- or off-pump or repeat (redo's) revascularisation procedures
2. Stable or unstable angina, including non ST-segment-elevation acute coronary syndrome (NSTE-ACS)
3. Age ≥ 18 years
4. Written informed consent

Exclusion Criteria:

1. Any concomitant cardiovascular procedure to CABG (i.e. valve, aortic or carotid surgery)
2. Acute ST-segment-elevation myocardial infarction (STEMI)
3. NSTE-ACS with cardiogenic shock warranting emergent salvage surgery within 12 hrs from hospital admission
4. History of atrial fibrillation or muscle disease (myopathy)
5. Current renal (creatinine>2x upper limit of normal (ULN), dialysis, kidney transplant) or hepatic dysfunction (AST/ALT>2x ULN, liver transplant or neoplasm)
6. Inability of oral drug intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2630 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiocerebral events (MACCE) within 30 days after CABG. | 30 days after Surgery
  Composite endpoint consisting of (1) all-cause mortality, (2) non-fatal myocardial infarction (MI) and (3) non-fatal cerebrovascular event (stroke or TIA).

SECONDARY OUTCOMES:
Major adverse cardiac events | 30 days after Surgery
  Composite outcome consisting cardiac mortality and non-fatal MI within 30 days after surgery.
Length of stay | within the first 15 days after surgery (plus or minus 5 days)
  Length of stay on intensive care unit (ICU) and hospital
Repeat coronary revascularisation | 30 days after surgery
  Repeat coronary revascularisation (PCI or CABG)
Mortality at 12 months | 12 months after surgery
  All-cause mortality at 12 months
Wound Infections | 30 days after surgery
  Surgical site wound infections.
Atrial fibrillation | within the first 15 days after surgery (plus or minus 5 days)
  New-onset postoperative atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Oliver J Liakopoulos, MD, PhD, Principal Investigator — University of Cologne
Locations (10):
- Germany (10):
  - Heart Center Freiburg-Bad Krozingen, Freiburg im Breisgau, Baden-Wurttemberg
  - Heart Center Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - University of Aachen, Aachen, North Rhine-Westphalia
  - Heart Center Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia
  - University of Bochum, Bochum, North Rhine-Westphalia
  - University of Bonn, Bonn, North Rhine-Westphalia
  - University of Cologne, Cologne, North Rhine-Westphalia
  - University of Essen, Essen, North Rhine-Westphalia
  - University of Muenster, Münster, North Rhine-Westphalia
  - Helios Heart Center Wuppertal, Wuppertal, North Rhine-Westphalia

REFERENCES:
- [Derived] Liakopoulos OJ, Kuhn EW, Hellmich M, Kuhr K, Krause P, Reuter H, Thurat M, Choi YH, Wahlers T; StaRT-CABG Investigators. Statin Recapture Therapy before Coronary Artery Bypass Grafting Trial: Rationale and study design of a multicenter, randomized, double-blinded controlled clinical trial. Am Heart J. 2015 Jul;170(1):46-54, 54.e1-2. doi: 10.1016/j.ahj.2015.04.015. Epub 2015 Apr 17. PMID 26093863
- See also: StaRT CABG Homepage — http://www.start-cabg.de